CLINICAL TRIAL: NCT01252875
Title: EVALUATION OF TWO SECONDARY CARE STRATEGIES AFTER STROKE OR TRANSIENT ISCHEMIC ATTACK (TIA): ACHEIVED TARGET LDL-C TO 100 mg/dL (+/- 10,mg/dL) OR LESS THAN 70 mg/dL.
Brief Title: Treat Stroke to Target
Acronym: TST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Pfizer (Industry); AstraZeneca (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P081244
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-06

CONDITIONS: Ischemic Stroke; Transient Ischemic Attack; Atherosclerotic Stenosis
Keywords: LDL-C; Cholesterol; Stroke; Transient ischemic attack; Statin; Lipid lowering therapy
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LDL-C to100 mg/dL (+/-10 mg/dL) (Other): Target : 100 mg/dL (+/-10 mg/dL):
  Patients recruited in this arm will receive statin +/-other lipid lowering therapy in order to reach a LDL-C concentration of 100 mg/dL(+/-10 mg/dL).
  Interventions: Procedure: Target : 100 mg/dL (+/-10 mg/dL)
- LDL-C < 70 mg/dL (Other): 70 mg/dL: Patients recruited in this arm will receive statin +/-other lipid lowering therapy in order to reach a LDL-C concentration of less than 70 mg/dL.
  Interventions: Procedure: 70 mg/dL

INTERVENTIONS:
Procedure: Target : 100 mg/dL (+/-10 mg/dL) — Statin +/- other lipid lowering therapy during 3 years, Target : LDL-C =100 mg/dL (+/-10 mg/dL), recording recurrent non fatal stroke, non fatal MI, and vascular death and others endpoints such as new onset diabetes, hemorrhagic strokes.
  Other Names: treat to target
  Arms: LDL-C to100 mg/dL (+/-10 mg/dL)
Procedure: 70 mg/dL — Statin +/-lipid lowering therapy during eight and a half years maximum, Target : LDL-C concentration of less than 70 mg/dL, recording recurrent of non fatal stroke, non fatal IM, and vascular death and others endpoints such as: new onset diabetes, hemorrhagic strokes.
  Other Names: treat to target
  Arms: LDL-C < 70 mg/dL

SUMMARY:
The aim of this study is the evaluation of two usual care strategies after stroke or TIA : achieved target LDL-C of 100 mg/dL (+/-10 mg/dL) or less than 70 mg/dL. Investigators will use the statin and titrate the dosage to achieve the target assigned by randomization in monotherapy or in combination with ezetimibe or other drugs.

The primary end-point is the occurrence of recurrent non fatal stroke, non fatal MI, and vascular death in each group.

3760 patients will be recruited and followed for eight and a half years maximum.

DETAILED DESCRIPTION:
The aim of this study is the evaluation of two usual care strategies after stroke or TIA : achieved target LDL-C of 100 mg/dL (+/-10 mg/dL) or less than 70 mg/dL. Investigators will use the statin and titrate the dosage to achieve the target assigned by randomization in monotherapy or in combination with ezetimibe or other drugs.

Inclusion criteria:

* Recent (less than 3 months) ischemic stroke As soon as possible after the event, once the neurologic deficit is stabilized (investigator judgment). These ischemic strokes include TIA with ischemic lesion documented by CT or MRI.
* Or recent TIA (less than 15 days) without documentation of ischemic lesion on CT/MR imaging. Must be limb weakness or aphasia lasting more than 10 min.
* And documented atherosclerotic stenosis in carotid artery (investigator judgment) (based on the results of Duplex echography, CTA, MRA or X ray- angiography), Or in the aortic arch (investigator judgment) (based on TEE or CTA), Or in other brain artery: vertebral, basilar or other intracranial artery (based on CTA, MRA, XRA), Or in coronary arteries (past history of acute coronary syndrome, coronary revascularization or positive coronary angiography)
* And statin treatment is indicated, following ANSM guidelines (French drug agency), age >18 years, rankin score ≤ 4, patient or a legal representative signs consent, patient is affiliated to social security system

Exclusion criteria :

* Ischemic stroke/TIA du to arterial dissection (investigator judgment)
* Cardiac source of embolism (e.g., mitral stenosis, endomyocardial fibrosis) without documented atherosclerotic stenosis : a patient with atrial fibrillation or a past history of recent myocardial infarction or calcified aortic stenosis can be randomized if he otherwise fulfils inclusion criteria
* Symptomatic hemorrhagic stroke : Presence of microbleeds on gradient echo imaging (T2*) is not an exclusion criteria. Hemorrhagic transformation of an ischemic stroke is not an exclusion criteria
* Uncontrolled hypertension (investigator judgment)
* LDL-C <100 mg/dL or patients for whom treatment intensification is impossible
* F/U impossible or bad observance anticipated.
* Co-morbid condition that may interfere with the F/U or with the evaluation of primary endpoint
* Participation to another clinical trial

The primary end-point is:

Recurrent ischemic stroke or stroke of undetermined origin, myocardial infarction, urgent coronary or carotid revascularization following new symptoms requiring hospitalization, and vascular death.

Secondary endpoints:

* Recurrent nonfatal ischemic stroke
* Nonfatal myocardial infarction
* Recurrent ischemic stroke, fatal or non
* Recurrent ischemic stroke or TIA
* Intracranial hemorrhage (intracerebral hemorrhage, subarachnoid hemorrhage, subdural hematoma)
* All stroke (ischemic or hemorrhagic)
* Any major coronary events (including fatal and nonfatal myocardial infarction)
* Any coronary heart disease end-point (myocardial infarction, hospitalization for acute corornary symptoms, coronary revascularization procedure)
* Any revascularisation procedure (coronary, carotid, or peripheral artery))
* Carotid artery revascularization procedure (urgent following new symptoms or elective)
* Vascular death (ischemic stroke or undetermined stroke, fatal myocardial infarction, other vascular deaths, sudden death, death of undetermined cause, i.e., without other cause documented such as cancer, infection, accident, suicide, etc…)
* All causes deaths
* Primary endpoint plus intracranial hemorrhage
* New onset diabetes

Hypothesis :

* Follow-up of three years
* Risk of primary end-point in the control group (Target LDL <100 mg/dL) : 4% per year (12 % at 36 months)
* 5% Alpha, 80% power, total number of subject is :
* 3068 patients with a RRR 25%
* 20% drop-out: 3760 patients (385 primary EP)

Study specifications Follow-up : eight and a half years Follow-up visit : every 6 months Number of centers (French Stroke Units, under the auspice of the French Neurovascular Society) : 60-100

Ancillary study As an ancillary study, 800 patients (400 in each arm in 4 centers) will participate in the TST-PLUS (Plaque Ultrasound Study), in which they will have three ultrasound examination (baseline, 1 year and 3 years) and baseline blood sampling. The primary endpoint of this substudy will be the rate of occurrence of new carotid plaque, with the hypothesis that Rate of plaque occurrence in the <100 mg/dL group will be 25% after 3 years (45% in EVA when atherosclerosis was present at baseline) RRR of plaque of 25% in the <70 mg/dL group Alpha 5%, power 80%

As an ancillary study, 1000 patients will participate in the TST-PGS (Pharmacogenetics) Study, in which they will have 1 blood sampling either at baseline or during one of the follow-up visits of TST. The aim of this study is to show that the benefit (risk of ischemic stroke, myocardial infarction, and vascular death) observed with a strategy of LDL-C <0.7 g / l compared to a strategy of LDL-C to 1 ± 0.1 g / l is higher in carriers of polymorphism 719Arg of the gene KIF-6 than non-carriers of this polymorphism.

ELIGIBILITY:
Inclusion Criteria:

* • Recent (less than 3 months) ischemic stroke
* As soon as possible after the event, once the neurologic deficit is stabilized (investigator judgment)
* These ischemic strokes include TIA with ischemic lesion documented by CT or MRI

  • Or recent TIA (less than 15 days)
* without documentation of ischemic lesion on CT/MR imaging
* Must be limb weakness or aphasia lasting more than 10 min

  • And documented atherosclerotic stenosis
* In carotid artery (investigator judgment) (based on the results of Duplex echography, CTA, MRA or X ray- angiography)
* Or in the aortic arch (investigator judgment) (based on TEE or CTA)
* Or in other brain artery: vertebral, basilar or other intracranial artery (based on CTA, MRA, XRA)
* Or in coronary arteries (past history of acute coronary syndrome, coronary revascularization or positive coronary angiography)

  • And
* Statin treatment is indicated, following ANSM guidelines (French drug agency)
* age >18 years
* rankin score ≤ 4
* patient or a legal representative signs consent
* Patient is affiliated to social security system

Exclusion Criteria:

* • Ischemic stroke/TIA du to
* arterial dissection (investigator judgment)
* Cardiac source of embolism (e.g., mitral stenosis, endomyocardial fibrosis) without documented atherosclerotic stenosis : a patient with atrial fibrillation or a past history of recent myocardial infarction or calcified aortic stenosis can be randomized if he otherwise fulfils inclusion criteria

  • Symptomatic hemorrhagic stroke
* Presence of microbleeds on gradient echo imaging (T2*) is not an exclusion criteria.
* Hemorrhagic transformation of an ischemic stroke is not an exclusion criteria

  * Uncontrolled hypertension (investigator judgment)
  * LDL-C <100 mg/dL or patients for whom treatment intensification is impossible
  * F/U impossible or bad observance anticipated.
  * Co-morbid condition that may interfere with the F/U or with the evaluation of primary endpoint
  * Participation to another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2873 (Actual)
Dates: Start 2010-03-15 (Actual); Primary Completion 2019-05-26 (Actual); Study Completion 2019-05-26 (Actual)

PRIMARY OUTCOMES:
recurrent ischemic stroke or stroke of undetermined origin, myocardial infarction, urgent coronary or carotid revascularization following new symptoms requiring hospitalization, and vascular death. | each 6 months
  recurrent ischemic stroke or stroke of undetermined origin, myocardial infarction, urgent coronary or carotid revascularization following new symptoms requiring hospitalization, and vascular death.

SECONDARY OUTCOMES:
Recurrent nonfatal ischemic stroke | each 6 months
  Recurrent nonfatal ischemic stroke
Nonfatal myocardial infarction | each 6 months
  Nonfatal myocardial infarction
Recurrent ischemic stroke, fatal or non | each 6 months
  Recurrent ischemic stroke, fatal or non
Recurrent ischemic stroke or TIA | each 6 months
  Recurrent ischemic stroke or TIA
Intracranial hemorrhage (intracerebral hemorrhage, subarachnoid hemorrhage, subdural hematoma) | each three weeks until target is not achieved then each 6 months
  Intracranial hemorrhage (intracerebral hemorrhage, subarachnoid hemorrhage, subdural hematoma)
All stroke (ischemic or hemorrhagic) | each three weeks until target is not achieved then each 6 months
  All stroke (ischemic or hemorrhagic)
Any major coronary events (including fatal and nonfatal myocardial infarction) | each 6 months
  Any major coronary events (including fatal and nonfatal myocardial infarction)
Any coronary heart disease end-point (myocardial infarction, hospitalization for acute corornary symptoms, coronary revascularization procedure) | each 6 months
  Any coronary heart disease end-point (myocardial infarction, hospitalization for acute corornary symptoms, coronary revascularization procedure)
Any revascularisation procedure (coronary, carotid, or peripheral artery)) | each 6 months
  Any revascularisation procedure (coronary, carotid, or peripheral artery))
Carotid artery revascularization procedure (urgent following new symptoms or elective) | each 6 months
  Carotid artery revascularization procedure (urgent following new symptoms or elective)
Vascular death (ischemic stroke or undetermined stroke, fatal myocardial infarction, other vascular deaths, sudden death, death of undetermined cause, i.e., without other cause documented such as cancer, infection, accident, suicide, etc…) | each 6 months
  Vascular death (ischemic stroke or undetermined stroke, fatal myocardial infarction, other vascular deaths, sudden death, death of undetermined cause, i.e., without other cause documented such as cancer, infection, accident, suicide, etc…)
All causes deaths | each 6 months
  All causes deaths
Primary endpoint plus intracranial hemorrhage | each 6 months
  Primary endpoint plus intracranial hemorrhage
New onset diabetes | each 6 months
  New onset diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Amarenco, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - BICHAT HOSPITAL Departement of Neurology, Paris
  - BICHAT HOSPITAL Department of neurology and stroke center, Paris

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Amarenco P, Lavallee PC, Kim JS, Labreuche J, Charles H, Giroud M, Lee BC, Mahagne MH, Meseguer E, Nighoghossian N, Steg PG, Vicaut E, Bruckert E; Treat Stroke to Target Investigators. More Than 50 Percent Reduction in LDL Cholesterol in Patients With Target LDL <70 mg/dL After a Stroke. Stroke. 2023 Aug;54(8):1993-2001. doi: 10.1161/STROKEAHA.123.042621. Epub 2023 Jun 28. PMID 37376989
- [Derived] Amarenco P, Kim JS, Labreuche J, Charles H, Giroud M, Lee BC, Lavallee PC, Mahagne MH, Meseguer E, Nighoghossian N, Steg PG, Vicaut E, Bruckert E; Treat Stroke to Target Investigators. Yield of Dual Therapy With Statin and Ezetimibe in the Treat Stroke to Target Trial. Stroke. 2022 Nov;53(11):3260-3267. doi: 10.1161/STROKEAHA.122.039728. Epub 2022 Sep 26. PMID 36154103
- [Derived] Amarenco P, Kim JS, Labreuche J, Charles H, Giroud M, Lavallee PC, Lee BC, Mahagne MH, Meseguer E, Nighoghossian N, Steg PG, Vicaut E, Bruckert E; Treat Stroke to Target Investigators*. Intracranial Hemorrhage in the TST Trial. Stroke. 2022 Feb;53(2):457-462. doi: 10.1161/STROKEAHA.121.035846. Epub 2021 Dec 29. PMID 34963300
- [Derived] Amarenco P, Kim JS, Labreuche J, Charles H, Giroud M, Lee BC, Lavallee PC, Mahagne MH, Meseguer E, Nighoghossian N, Steg PG, Vicaut E, Bruckert E; Treat Stroke to Target Investigators; Treat Stroke to Target investigators:. Impact of Lower Versus Higher LDL Cholesterol Targets on Cardiovascular Events After Ischemic Stroke in Patients With Diabetes. Diabetes. 2021 Aug;70(8):1807-1815. doi: 10.2337/db21-0302. Epub 2021 May 12. PMID 33980690
- [Derived] Amarenco P, Hobeanu C, Labreuche J, Charles H, Giroud M, Meseguer E, Lavallee PC, Gabriel Steg P, Vicaut E, Bruckert E, Touboul PJ. Carotid Atherosclerosis Evolution When Targeting a Low-Density Lipoprotein Cholesterol Concentration <70 mg/dL After an Ischemic Stroke of Atherosclerotic Origin. Circulation. 2020 Aug 25;142(8):748-757. doi: 10.1161/CIRCULATIONAHA.120.046774. Epub 2020 Jun 29. PMID 32594766
- [Derived] Amarenco P, Kim JS, Labreuche J, Charles H, Giroud M, Lee BC, Mahagne MH, Nighoghossian N, Gabriel Steg P, Vicaut E, Bruckert E; Treat Stroke to Target Investigators. Benefit of Targeting a LDL (Low-Density Lipoprotein) Cholesterol <70 mg/dL During 5 Years After Ischemic Stroke. Stroke. 2020 Apr;51(4):1231-1239. doi: 10.1161/STROKEAHA.119.028718. Epub 2020 Feb 20. PMID 32078484
- [Derived] Amarenco P, Kim JS, Labreuche J, Giroud M, Lee BC, Mahagne MH, Nighoghossian N, Simon T, Steg PG, Touboul PJ, Vicaut E, Yelles N, Bruckert E. Treat stroke to target trial design: First trial comparing two LDL targets in patients with atherothrombotic strokes. Eur Stroke J. 2019 Sep;4(3):271-280. doi: 10.1177/2396987319838100. Epub 2019 Mar 26. PMID 31984235
- [Derived] Amarenco P, Kim JS, Labreuche J, Charles H, Abtan J, Bejot Y, Cabrejo L, Cha JK, Ducrocq G, Giroud M, Guidoux C, Hobeanu C, Kim YJ, Lapergue B, Lavallee PC, Lee BC, Lee KB, Leys D, Mahagne MH, Meseguer E, Nighoghossian N, Pico F, Samson Y, Sibon I, Steg PG, Sung SM, Touboul PJ, Touze E, Varenne O, Vicaut E, Yelles N, Bruckert E; Treat Stroke to Target Investigators. A Comparison of Two LDL Cholesterol Targets after Ischemic Stroke. N Engl J Med. 2020 Jan 2;382(1):9. doi: 10.1056/NEJMoa1910355. Epub 2019 Nov 18. PMID 31738483